CLINICAL TRIAL: NCT05999591
Title: Effect of Post-Wash Total Motile Sperm Count on the Pregnancy Rate of Infertility Patients Undergoing Intrauterine Insemination
Brief Title: Total Motile Sperm Count and Pregnancy Rate From Intrauterine Insemination
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: OBGY-202308.01
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Insemination
Keywords: infertility; intrauterine insemination; post-wash total motile sperm count
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intrauterine insemination: Patients undergoing intrauterine insemination
  Interventions: Procedure: Intrauterine insemination

INTERVENTIONS:
Procedure: Intrauterine insemination — Transfer of sperm into the fallopian tube through a specialised cannula

SUMMARY:
Intrauterine insemination (IUI) is one of the most important infertility treatments. Infertility is failure to establish pregnancy (>12 months) with regularly unprotected sexual intercourse. Post-wash total motile sperm count (TMSC) vaguely defined as a predictor of IUI pregnancy rate. The minimum value required is also not clear. This study aimed to further define the relationship and determine the minimum recommended value to achieve a satisfactory IUI pregnancy rate.

Post-wash TMSC is predictive of IUI success. No optimal cut-off could be identified. In conclusion, post-wash TMSC is highly suggested as a quantitative predictor along with others in counseling and informed consent. The recommended threshold value is >3 x 106.

ELIGIBILITY:
Inclusion Criteria:

* post-wash total motile sperm count needed to be over 5 x 10^5

Exclusion Criteria:

* missing data on pregnancy outcome and missing medical records

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A group of patients undergoing intrauterine insemination for various causes of infertility at a tertiary fertility clinic
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-01-22 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | max 9 months
  Pregnancy number divided by number of IUI cycles

CONTACTS AND LOCATIONS:
Overall Officials: Hanom H Syam, M.D., Ph.D, Principal Investigator — Department of Obstetrics and Gynecology, Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Universitas Padjadjaran, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
anonymised patient data are available upon reasonable written request to the authors

REFERENCES:
- [Result] Miller DC, Hollenbeck BK, Smith GD, Randolph JF, Christman GM, Smith YR, Lebovic DI, Ohl DA. Processed total motile sperm count correlates with pregnancy outcome after intrauterine insemination. Urology. 2002 Sep;60(3):497-501. doi: 10.1016/s0090-4295(02)01773-9. PMID 12350496